CLINICAL TRIAL: NCT02888392
Title: The Effect of Zespri Green Kiwifruit on Digestive and Gut Health Functions: a Multi-country, Randomized, Cross-over Clinical Intervention
Brief Title: The Effect of Zespri Green Kiwifruit on Digestive and Gut Health Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zespri International Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HN1525
Record Dates: First submitted 2016-08-22; First posted 2016-09-05 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — alcohol acyltransferase, Actinidia; Psyllium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kiwifruit intervention (Experimental): 4 week intervention treatment with 2 fresh, whole green kiwifruit per day
  Interventions: Other: Kiwifruit
- Psyllium intervention (Active Comparator): 4 week intervention treatment with psyllium, matched for fibre content of 2 green kiwifruit / day for 4 weeks
  Interventions: Dietary Supplement: Psyllium

INTERVENTIONS:
Other: Kiwifruit — 2 green kiwifruit cultivar 'Hayward'
  Arms: Kiwifruit intervention
Dietary Supplement: Psyllium — Pysllium seed husk; ispaghula, isabgol, or psyllium, are portions of the seeds of the plant Plantago ovata, (genus Plantago), a native of India, Bangladesh and Pakistan. They are hygroscopic, which allows them to expand and become mucilaginous. Psyllium is a faecal bulking agent used to treat constipation. It absorbs liquid in the intestines, swells and forms a bulky soft stool that is easy to pass
  Other Names: Ispaghula, isabgol
  Arms: Psyllium intervention

SUMMARY:
The proposed study will primarily demonstrate the efficacy of kiwifruit as a food intervention for the relief of constipation and associated symptoms in functionally constipated adults, and those with IBS-C. Secondary measures will show the consumption of kiwifruit will result in improvements in gastro-intestinal discomfort levels of adults with IBS-C.

DETAILED DESCRIPTION:
The study is a randomised, single-blinded, cross-over design. Both target study populations (those with functional constipation, and the matched healthy control group) will complete the 16-week trial. Each study group will be randomly selected to either begin the first intervention period on the kiwifruit treatment or the psyllium treatment, and following the washout period will then receive the opposite treatment. Researchers and analysts will be blind as to as to the order of treatment individuals will receive. A dedicated treatment administrator will be assigned to provide the treatments to participants and liaise with them during the intervention phases.

All participants will be free living and required to maintain their normal dietary and lifestyle habits for the duration of the trial.

The primary outcome measure will be quantification of CSBM (complete spontaneous bowel movement). Secondary outcome measures will include additional stool frequency measures and other questionnaires.

ELIGIBILITY:
The study group will consist of 3 balanced groups of 20 subjects. A functionally constipated group (FC), an irritable bowel syndrome with constipation group (IBS-C), and a healthy control group (HC). The FC and IBS-C groups are the study population of interest to measure improvements in digestive comfort, and the HC will ensure no adverse events, confirming kiwifruit are suitable for consumption by the general healthy population.

All participants must fall within:

1. Adult (18-65 years). Females will be required to declare stage of menstrual cycle during the different trial phases.
2. BMI between 18-35 Screening questionnaires for participant selection, together with the sample ROME III FC/ IBS-C criteria screening questions are provided in Appendix C. This questionnaire enables potential participants to be screened for both FC and IBS-C, together with some "red flag" questions to further determine participant suitability.

Inclusion Criteria:

* The functionally constipated (FC) study participant group will be selected based on the following criteria:

  1. Presence of functional constipation according to ROME III diagnostic criteria*5b i. Must include two or more of the following:

     1. Straining during at least 25% of defecations
     2. Lumpy or hard stools in at least 25% of defecations
     3. Sensation of incomplete evacuation for at least 25% of defecations
     4. Sensation of anorectal obstruction/blockage for at least 25% of defecations
     5. Manual manoeuvres to facilitate at least 25% of defecations (e.g. digital evacuation, support of pelvic floor)
     6. Fewer than three defecations per week ii. Loose stools are rarely present without the use of laxatives iii. Insufficient criteria for irritable bowel syndrome * Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis
  2. Participants with IBS-C (mild). The diagnostic criteria * for Irritable Bowel Syndrome5a is:

     Recurrent abdominal pain or discomfort** at least 3 days per month in the last 3 months associated with 2 or more of the following:

     i. Improvement with defecation ii. Onset associated with a change in frequency of stool iii. Onset associated with a change in form (appearance of stool)

     * Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis

     ** Discomfort means an uncomfortable sensation not described as pain. In pathophysiology research and clinical trials, a pain/discomfort frequency of at least 2 days a week during screening evaluation for subject eligibility.

     IBS-C requires meeting the IBS criteria together with - hard or lumpy stools (Bristol Stool Form Scale 1-2) ≥ 25%, and loose or mushy stools ≤ 25% of bowel movements (Bristol Stool Form Scale 6-7).

     Exclusion Criteria:
* Potential participants will be excluded if they have any alarm features associated with bowel habit (recent changes in bowel habit (<3 months), rectal bleeding, weight loss, occult blood in stools, anaemia), anal fissures, bleeding haemorrhoids, and family history of GI cancer or IBD.

Chronic disease (cardiovascular, cancer, renal failure, previous gastrointestinal surgery (not including appendectomy or cholecystectomy), neurological conditions (e.g. multiple sclerosis, spinal chord injury, stroke).

All patients will be screened at recruitment for fasting blood glucose. Those with results ≥ 7.2 mmol/l will not be accepted into the trial.

Participants with diagnosed and stable conditions requiring the use of SSRI's (selective serotonin reuptake inhibitors), tricyclates, opiates or anti-inflammatories will be permitted into the trial on condition the medication has been in use continually and the condition has been stable for > 3 months. Similarly those with stable and controlled diabetes (> 3 months) will be permitted to participate.

Women who are pregnant, breastfeeding or planning a pregnancy in the 3 months post selection (trial period) will be excluded.

Potential participants with known kiwifruit or latex allergy will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Complete Spontaneous Bowel Motions | Total study duration per participant of 16 weeks. CSBM was assessed weekly from 2 week lead-in before baseline and every week through intervention 1, wash-out, intervention 2 and for a two week follow-up period .
  A spontaneous bowel motion not induced by rescue medication and associated with a sense of complete evacuation

SECONDARY OUTCOMES:
Daily Bowel Habit | Total study duration per participant of 16 weeks. Daily bowel habit was assessed daily from 2 week lead-in before baseline and every day through intervention 1, wash-out, intervention 2 and for a two week follow-up period .
  Frequency of bowel movements, ease of defaecation, stool form
Weekly Gastrointestinal Symptom Rating Scale (GSRS) | Total study duration per participant of 16 weeks. GSRS was assessed weekly from 2 week lead-in before baseline and every week through intervention 1, wash-out, intervention 2 and for a two week follow-up period .
  Gastrointestinal Symptom Rating Scale
Rome III | Total study duration per participant of 16 weeks. Rome III was assessed at the start of the study, 2 weeks later at baseline, and at the end of each study period i.e. after intervention 1, wash-out, intervention 2 and at the end of a 2 week follow up .
  Rome III questionnaire to establish patient group as Healthy, FC, or IBS-C
Irritable Bowel Syndrome Quality of Life (IBS-QoL) evaluation | Total study duration per participant of 16 weeks. Rome III was assessed at baseline, and at the end of each study period i.e. after intervention 1, wash-out, and the end of intervention 2.
  Validated quality of life questionnaire
Profile of Mood Score (POMS) | Total study duration per participant of 16 weeks. POMS was assessed at baseline, and at the end of each study period i.e. after intervention 1, wash-out, intervention 2 and at the end of a 2 week follow up .
  Validated mood score questionnaire
Irritable Bowel Syndrome severity score index (IBS-SSI) | IBS-SSI was completed once at enrollment
  Validated questionnaire to score severity of IBS to assign participants to correct group
3-day Food Diary | Total study duration per participant of 16 weeks. The food diary was done at baseline, and at the end of each study period i.e. after intervention 1, wash-out, and intervention 2
  3 day recall diet record to establish diet remains consistent throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barbara, MD, Principal Investigator — St. Orsola Hospital, University of Bologna
Locations (1):
- St. Orsola Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gearry R, Fukudo S, Barbara G, Kuhn-Sherlock B, Ansell J, Blatchford P, Eady S, Wallace A, Butts C, Cremon C, Barbaro MR, Pagano I, Okawa Y, Muratubaki T, Okamoto T, Fuda M, Endo Y, Kano M, Kanazawa M, Nakaya N, Nakaya K, Drummond L. Consumption of 2 Green Kiwifruits Daily Improves Constipation and Abdominal Comfort-Results of an International Multicenter Randomized Controlled Trial. Am J Gastroenterol. 2023 Jun 1;118(6):1058-1068. doi: 10.14309/ajg.0000000000002124. Epub 2022 Dec 20. PMID 36537785